CLINICAL TRIAL: NCT07035002
Title: Study on the Safety and Tolerability of PD-1 Knockout Tumor-infiltrating T Cells (TILs) in the Treatment of Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Prof., Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-570
Record Dates: First submitted 2025-06-07; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer (CRC); Tumor Infiltrating Lymphocytes; PD-1
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Low dose (Experimental): The dose of 5×10^8 PD-1 edited TILs per kg body weight will be transfused to 3 enrolled cases. If none of the 3 patients showed dose-limiting toxicity, the study would be proceeded and the dose would be escalated for group B. If one patient developed dose-limiting toxicity (DLT), another 3 patients with the same dose of group A would be added for expanded investigation. If there was lower than 1/6 of the patients in group A developed DLT, the study would be proceeded and the dose would be escalated for group B.
  Interventions: Biological: transfusion of 5×10^8 PD-1 knockout TILs per kg body weight
- Group B: Middle dose (Experimental): The dose of 1×10^9 PD-1 edited TILs per kg body weight will be transfused to 3 enrolled cases. If none of the 3 patients showed dose-limiting toxicity, the study would be proceeded and the dose would be escalated for group C. If one patient developed DLT, another 3 patients with the same dose of group B would be added for expanded investigation. If there was lower than 1/6 of the patients in group B developed DLT, the study would be proceeded and the dose would be escalated for group C. If there was more than 2/6 of the patients in group B developed DLT, the study would be proceeded with the dose would be dropped for group A.
  Interventions: Biological: transfusion of 1×10^9 PD-1 edited TILs per kg body weight
- Group C: High dose (Experimental): The dose of 2×10^9 PD-1 edited TILs per kg body weight will be transfused to 3 enrolled cases. If none of the 3 patients showed dose-limiting toxicity, the study would be proceeded for group D. If one patient developed DLT, another 3 patients with the same dose of group C would be added for expanded investigation. If there was more than 2/6 of the patients in group B developed DLT, the study would be proceeded with the dose would be dropped for group B.
  Interventions: Biological: transfusion of 2×10^9 PD-1 edited TILs per kg body weight
- Group D: Expanded investigation (Experimental): The highest dose of TILs without side effects in groups A, B and C would be transfused. In the case that there were no DLT in group A, B and C, there were total 11 cases in group D.
  Interventions: Biological: transfusion of maximum dose without side effects among group A, B and C

INTERVENTIONS:
Biological: transfusion of 5×10^8 PD-1 knockout TILs per kg body weight — Obtaining individual tumor tissue via surgery resection or biopsy, and then isolating TILs in the tumor under GMP conditions, and further using gene editing technology to knockout PD-1 to finally obtain gene-edited TILs-T cells, and transfusing them back to the patient.
  Arms: Group A: Low dose
Biological: transfusion of 1×10^9 PD-1 edited TILs per kg body weight — Obtaining individual tumor tissue via surgery resection or biopsy, and then isolating TILs in the tumor under GMP conditions, and further using gene editing technology to knockout PD-1 to finally obtain gene-edited TILs-T cells, and transfusing them back to the patient.
  Arms: Group B: Middle dose
Biological: transfusion of 2×10^9 PD-1 edited TILs per kg body weight — Obtaining individual tumor tissue via surgery resection or biopsy, and then isolating TILs in the tumor under GMP conditions, and further using gene editing technology to knockout PD-1 to finally obtain gene-edited TILs-T cells, and transfusing them back to the patient.
  Arms: Group C: High dose
Biological: transfusion of maximum dose without side effects among group A, B and C — Obtaining individual tumor tissue via surgery resection or biopsy, and then isolating TILs in the tumor under GMP conditions, and further using gene editing technology to knockout PD-1 to finally obtain gene-edited TILs-T cells, and transfusing them back to the patient.
  Arms: Group D: Expanded investigation

SUMMARY:
TIL from tumor tissue of advanced colorectal cancer patients were cultured, modified and expanded in vitro, and then transfused back to the patients after quality control. The safety and efficacy of the treatment were investigated. The fundamental cause of oncogenesis lies in the accumulation of gene mutations. A large number of gene mutations in tumor cells lead to changes in the encoded amino acid sequence, resulting in the production of tumor-specific proteins. Human T cells recognize tumor-specific peptides (tumor neoantigens) that are presented on the MHC molecules on the surface of tumor cells, leading to T cell enrichment within the tumor. However, due to the immunosuppressive effect of tumors through various ways, the enriched T cells in tumors cannot effectively kill tumor cells. One of the most common examples is that tumors up-regulate the expression of immune checkpoint protein PD-L1, which binds to PD-1 on the surface of T cells and inhibits T cell function. Therefore, in this study, we will obtain tumor tissue via surgery resection or biopsy, and then isolate TIL cells in the tumor under GMP conditions, and further use gene editing technology to knockout PD-1, the obtained gene-edited T cells will have the characteristics of specific recognition of tumor cells, but not sensitive to the immunosuppressive function of tumor cells, so as to achieve the therapeutic effect on tumor patients.

DETAILED DESCRIPTION:
Study name: Study on the safety and tolerability of PD-1 gene knockout tumor-infiltrating T cells (TIL) in the treatment of advanced colorectal cancer.

About the study: TIL from tumor tissue of advanced colorectal cancer patients were cultured, modified and expanded in vitro, and then transfused back to the patients after quality control. The safety and efficacy of the treatment were investigated. The fundamental cause of oncogenesis lies in the accumulation of gene mutations. A large number of gene mutations in tumor cells lead to changes in the encoded amino acid sequence, resulting in the production of tumor-specific proteins. Human T cells recognize tumor-specific peptides (tumor neoantigens) that are presented on the MHC molecules on the surface of tumor cells, leading to T cell enrichment within the tumor. However, due to the immunosuppressive effect of tumors through various ways, the enriched T cells in tumors cannot effectively kill tumor cells. One of the most common examples is that tumors up-regulate the expression of immune checkpoint protein PD-L1, which binds to PD-1 on the surface of T cells and inhibits T cell function. Therefore, in this study, we will obtain tumor tissue via surgery resection or biopsy, and then isolate TIL cells in the tumor under GMP conditions, and further use gene editing technology to knockout PD-1, the obtained gene-edited T cells will have the characteristics of specific recognition of tumor cells, but not sensitive to the immunosuppressive function of tumor cells, so as to achieve the therapeutic effect on tumor patients.

Objectives of the study:

Primary objective: To evaluate the safety and tolerability of PD-1 knockout TILs transfer treatment.

Secondary objectives: Objective response rate (ORR) and overall survival (OS) of PD-1 knockout TILs transfer treatment.

Subjects: The subjects were patients with advanced colorectal cancer confirmed by histology or cytology, who were not eligible to standard treatment at this stage. There were no restrictions on sex and region of origin, and patients volunteered to receive surgery or biopsy to obtain tumor tissue for TILs preparation. Aged ≥18 and ≤70 years old. At least one tumor lesion that could be evaluated according to RECIST, version 1.1. ECOG score was 0 or 1. Adequate bone marrow and organ function. A total of 20 patients were enrolled. The expected survival time of the enrolled patients was no less than 6 months.

Research setting/location: Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine Study intervention: TILs were isolated from tumor tissue and infused back into patients after PD-1 knockout and expanded culturing. The patients were treated with cyclophosphamide and fludarabine before TILs transfusion.

The evaluation of efficacy included: the concentration of cytokines in blood, the number and duration of TILs in blood, adverse complications, evaluations of tumor size based on RESIST v1.1(by B-ultrasound, CT or MRI), tumor biomarkers, tumor related ctDNA.

Study Duration: The overall study duration was 24 months, including the time from the recruitment of the first patient to the completion of the data analysis of the last patient.

Duration of subject participation: Each enrolled patient was followed up for 12 months after completion of the TILs transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced colorectal cancer confirmed by histology or cytology, who were not eligible to standard treatment at this stage.
* Patients volunteered to receive surgery or biopsy to obtain tumor tissue for TILs preparation.
* Aged ≥18 and ≤70 years old.
* At least one tumor lesion that could be evaluated according to RECIST, version 1.1.
* ECOG score was 0 or 1.
* Adequate bone marrow and organ function.
* The expected survival time of the enrolled patients was no less than 6 months.

Exclusion Criteria:

* Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, traditional Chinese medicine with anti-tumor indications and other anti-tumor treatments within 2 weeks before sampling, except the following:

  1. Nitrosourea or mitomycin C within 6 weeks before surgery;
  2. Oral fluorouracils and small molecule targeted drugs for 1 week before surgery.
* Received other unmarketed investigational drug or treatment within 4 weeks before sampling;
* Had undergone major organ surgery (excluding needle biopsy) within 4 weeks before sampling or had significant lesions Trauma, or the need for elective surgery during the trial;
* Received systemic glucocorticoid (prednisone >10mg/ day or equivalent dose) or other immunosuppressive therapy within 14 days before sampling; Treatment with topical, ocular, intra-articular, nasal, and inhaled glucocorticoids was excluded. Short-term prophylaxis with glucocorticoids (e.g., to prevent contrast allergy)
* Use of immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferin, etc., within 14 days before sampling;
* Administration of live attenuated vaccine within 4 weeks before sampling;
* The toxicity of previous antineoplastic therapy has not recovered to CTCAE 5.0 grade ≤1 (except for alopecia and other researchers who judged that there was no safety risk);
* Patients with symptomatic central nervous system or leptomeningeal metastases or other evidence of uncontrolled central nervous system or leptomeningeal metastases as judged by the investigator to be ineligible for enrollment;
* Patients with active infection within 1 week before sampling and currently requiring systemic anti-infective treatment;
* A history of immunodeficiency, including positive HIV antibody test;
* Hepatitis B (HBsAg positive and/or hepatitis C (anti-HCV positive) and/or treponema pallidum antibody positive;
* Patients with current interstitial lung disease;
* Has a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree II-III atrioventricular block, etc.
  2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first dose of dose.
  3. New York Heart Association (NYHA) functional class ≥II or left ventricular ejection fraction (LVEF) <50%, or structural heart disease at high risk as judged by other investigators;
  4. clinically uncontrolled hypertension.
* Patients with active or previous autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), excluding patients with clinically stable autoimmune thyroid diseases and well-controlled type I diabetes;
* Received immunotherapy with grade ≥ 3 irAE;
* Clinically uncontrollable serous cavity effusion, which was judged by the investigator as not suitable for enrollment;
* Known alcohol or drug dependence;
* Persons with mental disorders or poor compliance;
* Pregnant or lactating women;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance as the highest dose without side effects | From enrollment to the end of follow up at 12 months
  Without the following side effects from each drug:
  1. Cyclophosphamide: suppression of bone marrow, nausea, mucositis, rash, hemorrhagic cystitis, myocardial injury, alopecia, infertility, nausea and vomiting, syndrome of abnormal secretion of antidiuretic hormone (SIADH).
  2. Fludarabine: myelosuppression, fever, chills, nausea and vomiting, malaism, fatigue, anorexia, weakness, neurotoxicity and interstitial pneumonia.
  3. General antibiotics: anaphylaxis, renal insufficiency, nausea, vomiting, liver damage, myelosuppression, photosensitivity.
  4. High-dose IL-2: High-dose IL-2 has a variety of side effects. Since the most common side effects are due to the adjuvant drugs used in the treatment, the main interventions we will take to reduce the occurrence of serious side effects include: timely monitoring of patients after drug administration and cell infusion, providing adequate clinical support measures and complete first aid protocols, and adjusting according to patients' response.
Safety as severe treatment related complications | From enrollment to the end of follow up at 12 months
  The rates of complications occurred, including :
  1. Cyclophosphamide: suppression of bone marrow, nausea, mucositis, rash, hemorrhagic cystitis, myocardial injury, alopecia, infertility, nausea and vomiting, syndrome of abnormal SIADH.
  2. Fludarabine: myelosuppression, fever, chills, nausea and vomiting, malaism, fatigue, anorexia, weakness, neurotoxicity and interstitial pneumonia.
  3. General antibiotics: anaphylaxis, renal insufficiency, nausea, vomiting, liver damage, myelosuppression, photosensitivity.
  4. High-dose IL-2: High-dose IL-2 has a variety of side effects. Since the most common side effects are due to the adjuvant drugs used in the treatment, the main interventions we will take to reduce the occurrence of serious side effects include: timely monitoring of patients after drug administration and cell infusion, providing adequate clinical support measures and complete first aid protocols, and adjusting in real time according to patients' response.

SECONDARY OUTCOMES:
Objective response rate | From enrollment to the end of follow up at 12 months
Overall survival | From enrollment to the end of follow up at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, None Selected, China

IPD SHARING:
Plan to Share IPD: No